CLINICAL TRIAL: NCT03199976
Title: Efficacy of Intermittent Tiotropium in Early Childhood Wheezing
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Subjects in the Salbutamol group discontinued the intervention more often due to troublesome respiratory symptoms
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Anne Kotaniemi-Syrjänen, MD, PhD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TFS01; 2015-002985-22 (EudraCT Number)
Record Dates: First submitted 2017-06-26; First posted 2017-06-27 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Wheezy Bronchitis; Asthmatic Bronchitis; Wheezing; Obstruction Airway
Keywords: wheeze; shortness of breath
MeSH Terms: conditions — Bronchiolitis; Respiratory Sounds; Airway Obstruction; Dyspnea | interventions — Tiotropium Bromide; Fluticasone; Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tiotropium Bromide & Salbutamol (Experimental): Inhaled Tiotropium Bromide 5 µg once a day, beginning at the onset of an upper respiratory tract infection and continuing for 7 to 14 days as needed, and inhaled Salbutamol 0.2 mg 4 to 6 times a day as needed for wheeze and shortness of breath
  Interventions: Drug: Tiotropium Bromide; Drug: Salbutamol
- Fluticasone Propionate & Salbutamol (Active Comparator): Inhaled Fluticasone Propionate 125 µg twice a day, beginning at the onset of an upper respiratory tract infection and continuing for 7 to 14 days as needed, and inhaled Salbutamol 0.2 mg 4 to 6 times a day as needed for wheeze and shortness of breath
  Interventions: Drug: Fluticasone Propionate; Drug: Salbutamol
- Salbutamol (Active Comparator): Inhaled Salbutamol 0.2 mg 4 to 6 times a day as needed for wheeze and shortness of breath
  Interventions: Drug: Salbutamol

INTERVENTIONS:
Drug: Tiotropium Bromide — Tiotropium Bromide 2.5 µg/dose inhaled aerosol
  Other Names: Spiriva Respimat
  Arms: Tiotropium Bromide & Salbutamol
Drug: Fluticasone Propionate — Fluticasone Propionate 125 µg/dose inhaled aerosol
  Other Names: Flixotide Evohaler
  Arms: Fluticasone Propionate & Salbutamol
Drug: Salbutamol — Salbutamol 0.1 mg/dose inhaled aerosol
  Other Names: Ventoline Evohaler

SUMMARY:
This study evaluates the effect of intermittent tiotropium bromide and salbutamol as needed versus intermittent fluticasone propionate and salbutamol as needed, or solely, salbutamol as needed on episode-free days in infants and toddlers with recurrent episodes of wheeze and/or shortness of breath.

DETAILED DESCRIPTION:
Up to 30% of all children suffer from episodic wheeze or shortness of breath, i.e. asthmatic bronchitis, during the first three years of life. The condition is usually induced by viral respiratory infections, and short-acting beta-agonists are recommended as a monotherapy for symptoms unless there are at least four physician-confirmed episodes of wheeze or shortness of breath, or three episodes plus asthma risk factors. There is a current need for new therapeutic agents to treat asthmatic bronchitis in young children.

In viral-induced wheeze, increased parasympathetic nerve activity results in increased acetylcholine release from nerve endings. Tiotropium bromide, an inhaled anticholinergic agent, prevents the acetylcholine function and achieves mild bronchodilatation and decrease in mucus secretion from the submucosal glands.

The aim of the study is to find out the effect of intermittent tiotropium bromide and salbutamol as needed versus intermittent fluticasone propionate and salbutamol as needed, or solely, salbutamol as needed on episode-free days in infants and toddlers with recurrent episodes of wheeze and/or shortness of breath. Episode-free days are defined as those days during which there are no symptoms of wheeze and/or shortness of breath, no unscheduled medical visits for wheeze and/or shortness of breath, and no use of rescue or supplementary controller medications.

ELIGIBILITY:
Inclusion Criteria:

1. Children at the age of 6 to 35 months.
2. Two to four physician-confirmed episodes of wheeze and/or shortness of breath.
3. Parents/legal representatives with sufficient written and spoken skills in Finnish language.

Exclusion Criteria:

1. Birth before 36th week of gestation.
2. Suspected/diagnosed chronic parenchymal lung disease or a structural airway defect, or a history of thoracotomy with pulmonary resection.
3. A history of congenital or acquired heart disease, including any unstable or life-threatening cardiac arrhythmia.
4. Constipation with a need of regular medication, or a diagnosed/suspected structural defect in the gastrointestinal tract.
5. A history of malignancy, or other significant chronic disorder, disease, or defect.

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2016-04-20 (Actual); Primary Completion 2020-11-18 (Actual); Study Completion 2020-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mika J Mäkelä, Professor, Study Director — Skin and Allergy Hospital, Helsinki University Hospital, Helsinki, Finland
Locations (1):
- Skin and Allergy Hospital, Helsinki University Hospital, Helsinki, Finland, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No
Deidentified individual participant data will not be made available.

REFERENCES:
- [Derived] Kotaniemi-Syrjanen A, Klemola T, Koponen P, Jauhola O, Aito H, Malmstrom K, Malmberg LP, Rahiala E, Sarna S, Pelkonen AS, Makela MJ. Intermittent Tiotropium Bromide for Episodic Wheezing: A Randomized Trial. Pediatrics. 2022 Sep 1;150(3):e2021055860. doi: 10.1542/peds.2021-055860. PMID 35942814

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tiotropium Bromide & Salbutamol | Fluticasone Propionate & Salbutamol | Salbutamol
Started | 27 | 25 | 28
Completed | 23 | 18 | 14
Not Completed | 4 | 7 | 14
Not completed — Lack of Efficacy | 3 | 6 | 13
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tiotropium Bromide & Salbutamol | Fluticasone Propionate & Salbutamol | Salbutamol | Total
Number analyzed (Participants) | 27 | 25 | 28 | 80
Age, Continuous [Mean (Standard Deviation); unit: months] | 21.4 (7.0) | 20.0 (6.8) | 22.1 (6.0) | 21.2 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 10 | 28
  Male | 18 | 16 | 18 | 52
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Finland | 27 | 25 | 28 | 80

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Episode-Free Days
Description: Effect on the episode-free days defined as the days during which there are no symptoms of wheeze and/or shortness of breath, no unscheduled medical visits for wheeze and/or shortness of breath, and no use of rescue or supplementary controller medications.
Time Frame: Up to 48 weeks
Population: Only those children with diary data available were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: percentage of episode-free days
Arm/Group | Tiotropium Bromide & Salbutamol | Fluticasone Propionate & Salbutamol | Salbutamol
Number analyzed (Participants) | 26 | 25 | 26
percentage of episode-free days | 97 [93 to 99] | 87 [78 to 93] | 88 [79 to 95]
Statistical Analysis 1: Comparison: Tiotropium Bromide & Salbutamol vs Fluticasone Propionate & Salbutamol vs Salbutamol; Test type: Superiority; p < 0.01, Wilcoxon (Mann-Whitney) — Bonferroni correction was applied in pairwise analyses

2. Secondary Outcome: Number of Participants With Unscheduled Physician Visits
Description: Effect on the number of unscheduled physician visits for episodes of wheeze and/or shortness of breath.
Time Frame: Up to 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Tiotropium Bromide & Salbutamol | Fluticasone Propionate & Salbutamol | Salbutamol
Number analyzed (Participants) | 27 | 25 | 28
Participants | 10 | 10 | 14
Statistical Analysis 1: Comparison: Tiotropium Bromide & Salbutamol vs Fluticasone Propionate & Salbutamol vs Salbutamol; Test type: Superiority; p = 0.595, Chi-squared

3. Secondary Outcome: Percentage of Days Participants Needed Rescue Medication
Description: Effect of the treatment on the need for bronchochilative and/or supplementary controller medication.
Time Frame: Up to 48 weeks
Population: Only patients with diary data available were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: percentage of days
Arm/Group | Tiotropium Bromide & Salbutamol | Fluticasone Propionate & Salbutamol | Salbutamol
Number analyzed (Participants) | 26 | 25 | 26
percentage of days | 2 [0 to 7] | 13 [6 to 21] | 12 [6 to 20]
Statistical Analysis 1: Comparison: Tiotropium Bromide & Salbutamol vs Fluticasone Propionate & Salbutamol vs Salbutamol; Test type: Superiority; p < 0.01, Wilcoxon (Mann-Whitney) — Bonferroni correction was applied in pairwise analyses

4. Secondary Outcome: Number of Participants With Adverse Events
Description: Occurrence of adverse events in treatment groups.
Time Frame: Up to 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Tiotropium Bromide & Salbutamol | Fluticasone Propionate & Salbutamol | Salbutamol
Number analyzed (Participants) | 27 | 25 | 28
Participants | 23 | 25 | 26
Statistical Analysis 1: Comparison: Tiotropium Bromide & Salbutamol vs Fluticasone Propionate & Salbutamol vs Salbutamol; Test type: Superiority; p < 0.05, Chi-squared

ADVERSE EVENTS:
Time Frame: 48 weeks
Arm/Group | Tiotropium Bromide & Salbutamol | Fluticasone Propionate & Salbutamol | Salbutamol
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/25 | 0/28
Serious Adverse Events (participants affected / at risk) | 4/27 | 3/25 | 3/28
Other Adverse Events (participants affected / at risk) | 19/27 | 22/25 | 23/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tiotropium Bromide & Salbutamol (N=27) | Fluticasone Propionate & Salbutamol (N=25) | Salbutamol (N=28)
Wheezy bronchitis and pneumonia (Infections and infestations) | 0 | 0 | 1
Wheezy bronchitis and laryngitis (Infections and infestations) | 0 | 1 | 0
Wheezy bronchitis and anaphylaxis to cashew (Infections and infestations) | 0 | 1 | 0
Wheezy bronchitis (Infections and infestations) | 3 | 1 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0
Enteritis (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tiotropium Bromide & Salbutamol (N=27) | Fluticasone Propionate & Salbutamol (N=25) | Salbutamol (N=28)
Otitis media (Infections and infestations) | 16 | 9 | 12
Upper respiratory tract infection (Infections and infestations) | 13 | 13 | 9
Wheezy bronchitis (Infections and infestations) | 7 | 7 | 12
Conjunctivitis (Infections and infestations) | 4 | 1 | 7
Enteritis (Infections and infestations) | 3 | 3 | 2
Minor trauma (Injury, poisoning and procedural complications) | 2 | 3 | 2
Eczema (Skin and subcutaneous tissue disorders) | 1 | 3 | 1
Exanthema (Skin and subcutaneous tissue disorders) | 1 | 2 | 2
Tonsillitis (Infections and infestations) | 1 | 1 | 3
Pharyngitis (Infections and infestations) | 2 | 0 | 2

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/76/NCT03199976/Prot_SAP_000.pdf